CLINICAL TRIAL: NCT00928733
Title: The Effect of Ethanol on Intestinal Permeability and Integrity in Healthy Individuals
Brief Title: Effects of Ethanol on Intestinal Permeability and Integrity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 09-3-026
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: Permeability; tight junctions; cytokines; inflammatory bowel diseases; The effect of alcohol on the intestinal permeability may have major consequences on health.; It's generally accepted that an increased intestinal permeability in alcoholic subjects lead; to translocation of bacterial endotoxins from the gut lumen into the portal vein and then to the liver.; In the liver, endotoxins trigger the immune system and activate the resident macrophages, Kupffer cells.; Activation of Kupffer cells leads to production of chemokines (IL-8) and; proinflammatory cytokines (IL-1, TNFα),resulting in hepatocytes damage, inflammation, fibrosis and finally cirrhosis.
MeSH Terms: conditions — Inflammatory Bowel Diseases; Inflammation; Fibrosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- alcohol (Experimental): Intraduodenal infusion of ethanol
  Interventions: Device: Gastroduodenoscopy- Intraduodenal intubation
- Ethanol (Other)
  Interventions: Device: Gastroduodenoscopy- Intraduodenal intubation
- Placebo (Experimental): Intraduodenal infusion of tap water
  Interventions: Device: Gastroduodenoscopy- Intraduodenal intubation

INTERVENTIONS:
Device: Gastroduodenoscopy- Intraduodenal intubation — 20 g ethanol diluted up to 10% in tap water

SUMMARY:
Alcohol consumption is a major health problem worldwide. It affects all systems of the body especially the gastrointestinal tract. Acute or chronic alcohol consumption has deleterious effects on the gastrointestinal mucosa vary from increased intestinal permeability, structural changes to sever destruction of the epithelial lining cells. Human data are still limited and most of the studies were performed in chronic alcohol abusers.

The investigators hypothesize that moderate alcohol drinking also may increase small intestinal permeability and contribute to the subsequent disruption of the tight junction complex. This study may provide more insight into the effects of moderate alcohol drinking on the small intestinal permeability.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Male gender to avoid the gender-related differences in ethanol metabolism.
* Between 18-45 years to avoid age-related changes in ethanol metabolism39.
* Normal medical history and physical examination.
* Normal liver function tests (i.e. ALT, AST, and γGT) according to the reference values for normal ranges of the liver enzymes at the laboratory of clinical chemistry of the Maastricht University Medical Center.
* Caucasian ethnicity.
* BMI=18 - 30 kg/m2.

Exclusion Criteria:

* History of gastro-intestinal disorders or abdominal surgery.
* History of alcohol abuse or current excessive alcohol consumption (> 2 alcoholic beverages per day or > 14 alcoholic beverages per week)40.
* Recent or chronic medications that may interact with ethanol metabolism or intestinal permeability i.e., NSAIDs, benzodiazepines and antidepressants.
* Smoking.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2009-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To assess intestinal permeability by means of sugar permeability testing after intraduodenal administration of ethanol. | 2 years

SECONDARY OUTCOMES:
To assess tight junctions structure and proteins in biopsy specimens after intraduodenal administration of ethanol. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: A Masclee, MD PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Draper LR, Gyure LA, Hall JG, Robertson D. Effect of alcohol on the integrity of the intestinal epithelium. Gut. 1983 May;24(5):399-404. doi: 10.1136/gut.24.5.399. PMID 6840613
- [Background] Hirsch S, Chaves G, Gotteland M, de la Maza P, Petermann M, Barrera P, Bunout D. [Intestinal permeability in alcoholic patients without liver damage]. Rev Med Chil. 1997 Jun;125(6):653-8. Spanish. PMID 9515283
- [Background] Basuroy S, Sheth P, Mansbach CM, Rao RK. Acetaldehyde disrupts tight junctions and adherens junctions in human colonic mucosa: protection by EGF and L-glutamine. Am J Physiol Gastrointest Liver Physiol. 2005 Aug;289(2):G367-75. doi: 10.1152/ajpgi.00464.2004. Epub 2005 Feb 17. PMID 15718285
- [Result] Elamin E, Masclee A, Troost F, Pieters HJ, Keszthelyi D, Aleksa K, Dekker J, Jonkers D. Ethanol impairs intestinal barrier function in humans through mitogen activated protein kinase signaling: a combined in vivo and in vitro approach. PLoS One. 2014 Sep 16;9(9):e107421. doi: 10.1371/journal.pone.0107421. eCollection 2014. PMID 25226407
- See also: Increased intestinal permeability — http://www.leakygut.co.uk/